CLINICAL TRIAL: NCT04375163
Title: Effects of Massage Between Sets of an Intense Isokinetic Exercise- Protocol of Knee Extensors in Tae Kwon Do Athletes on Knee Range of Motion, Thigh Circumference and Delayed Onset Muscle Soreness
Brief Title: Effects of Massage Between Sets of an Intense Isokinetic Exercise- Protocol of Knee Extensors in Tae Kwon Do Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Evaggelos Sykaras, Associate Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-9/2020
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-05

CONDITIONS: Athletic Performance
Keywords: sport massage; delayed onset muscle soreness; muscles recovery; continuous concentric eccentric exercise

STUDY DESIGN:
Intervention Model Description: 26 Tae Kwon Do athletes performed a vigorous exercise program on the isokinetic dynamometer twice in a period of 10 days, each time on a different extremity. In this way two groups of 26 individuals each were created, with the same individuals alternating. In the massage group (ME) a sport massage was applied between the sets while in the control group (NME) the break was passive. knee flexion and extension ROM, thigh circumference, and creatine kinase (CK) levels in blood plasma were measured before and after each test while L-DOMS was measured 24, 48, 72 and 96 hours after the exercise.
Who Masked: Outcomes Assessor
Masking Description: Assessor-blind randomized control trial. A masked assessor conducted the measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage group (ME) (Experimental): A sport massage was applied between the sets of an intense isokinetic exercise protocol for knee extensor muscles
  Interventions: Other: Isokinetic intense exercise protocol; Other: Massage treatment
- Control (Active Comparator): the break between the sets of an intense isokinetic exercise protocol for knee extensor muscles was passive
  Interventions: Other: Isokinetic intense exercise protocol

INTERVENTIONS:
Other: Isokinetic intense exercise protocol — The isokinetic protocol included 6 sets of 10 maximum efforts at 60 °/s of one leg with a 2-minute break between the sets.
Other: Massage treatment — Massage consisted of stroking (30") and petrissage (50") for muscle relaxation, then friction (10"), pincement and clapping (30") to prepare muscles for the next set.
  Arms: Massage group (ME)

SUMMARY:
26 Tae Kwon Do athletes performed a vigorous exercise program on the isokinetic dynamometer twice in a period of 10 days, each time on a different extremity. In this way two groups of 26 individuals each were created, with the same individuals alternating. In the massage group (MG) a sport massage was applied between the sets while in the control group (NMG) the break was passive.

DETAILED DESCRIPTION:
Objective: Τo investigate the effects of massage in athletic performance when applied during intervals of an intense isokinetic exercise protocol for knee extensor muscles.

Design: Randomized Controlled Trial. Participants: 26 Tae Kwon Do athletes performed a vigorous exercise program on the isokinetic dynamometer twice in a period of 10 days, each time on a different extremity. In this way two groups of 26 individuals each were created, with the same individuals alternating. In the massage group (MG) a sport massage was applied between the sets while in the control group (CG) the break was passive.

Main Outcome Measures: knee flexion and extension ROM, thigh circumference, and creatine kinase (CK) levels in blood plasma were measured before and after each test while L-DOMS was measured 24, 48, 72 and 96 hours after the exercise.

ELIGIBILITY:
Inclusion Criteria:

* Professional athletes
* Age range between 18-25.

Exclusion Criteria:

* Conduction of any strengthening exercises on the day before the tests
* Musculoskeletal injury during the last six months
* Background of knee trauma and/or surgery

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Changes in Active Knee Range of Motion (ROM) | day 1: pre-treatment, after- treatment, day: 10 pre-treatment, after- treatment
  The ROM of knee flexion and extension was measured before and after the exercise program application in both trials. In particular, the active knee extension was measured in the supine position and the active flexion in the prone position using a universal type goniometer.
Changes in creatine kinase (CK) levels in blood plasma | day 1: pre-treatment, after- treatment, day: 10 pre-treatment, after- treatment
  Blood samples were taken before and 24 hours after the isokinetic protocol to determine whether the exercise program caused fatigue and muscle damage. The blood sample was analyzed to determine CK activity levels in blood plasma using an in-vitro quantitative assay followed by a photometer
Changes in thigh circumference | day 1: pre-treatment, after- treatment, day: 10 pre-treatment, after- treatment
  The circumference of the thigh was measured with a tape measure before the test and after the exercise program at fixed spots at a distance of 10 and 20 cm from the center of the patella
Changes in Delayed Onset Muscle Soreness (DOMS) | day 1: 24, 48, 72 and 96 hours after-exercise, day 10: 24, 48, 72 and 96 hours after-exercise
  The DOMS measurement for the lower extremities (L-DOMS) was performed with the VAS scale 24, 48, 72 and 96 hours after the completion of the program. The VAS scale was tentative where 1 corresponded to "no soreness" and 10 to "very, very sore". The L-DOMS was assessed according to Doma et al1,22 and according to Jakeman et al, through questioning after they completed a body weight squat until their knees were flexed to approximately 90°

SECONDARY OUTCOMES:
Changes in concentric and eccentric torque | day 1: pre-treatment
  During the baseline testing session, the maximum concentric and eccentric torque of knee extensors at 60 °/s was measured with the Cybex Norm.The participant then sat in the armchair of the isokinetic dynamometer with his arms crossed in the chest. Two crossed straps held the torso firmly on the back of the armchair and a belt with an additional strap held the pelvis still. Each participant performed 3 maximal efforts with each leg and the best of the 3 efforts was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Evaggelos Sykaras, Study Director — Department of Physical Education and Sports Sciences
Locations (1):
- Department of Physical Education and Sports Sciences, Thessaloniki, Central Makedonia, Greece

IPD SHARING:
Plan to Share IPD: No